CLINICAL TRIAL: NCT05927480
Title: Audio Distraction for Traction Pin Placement: A Randomized Controlled Trial
Brief Title: Audio Distraction for Traction Pin Placement
Acronym: ADTPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Jackson Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A17-285
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-05

CONDITIONS: Lower Extremity Fracture
Keywords: Skeletal Traction; Audio Distraction

STUDY DESIGN:
Intervention Model Description: There are two treatment arms. Each undergo traction pin placement, but one arm is provided headphones with music while the other is not offered anything.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio Distraction (Experimental): Those included in this study and randomized into the treatment arm will be given an mp3 device and headphones to listen to genre of music of their choosing in addition to be treated to the routine care with the skeletal traction pin.
  Interventions: Behavioral: Audio distraction
- Control (No Intervention): Those randomized into this arm will receive the current routine care which is treatment with a skeletal traction pin and no audio distraction.

INTERVENTIONS:
Behavioral: Audio distraction — Music on an mp3 player will be provided to the patient for them to listen to while having the traction pin placed.
  Arms: Audio Distraction

SUMMARY:
Traction pin placement is a common way to temporarily manage femur fractures and unstable acetabular fractures while awaiting surgery. Skeletal traction is thought to reduce patient discomfort by improving fracture alignment as well as relaxing muscle spasm pain felt from the broken bone by stretching out the leg. Skeletal traction may also help prevent articular surface damage in the hip by decreasing joint pressure. Despite the benefits of skeletal traction, insertion of the traction pin can be a painful and unpleasant experience for the patient. Our study hopes to see if listening to music with headphones during insertion of the traction pin decrease patient pain and anxiety.

DETAILED DESCRIPTION:
Given that skeletal traction is the current standard of care at our institution; our study will focus on the use of audio distraction during placement of skeletal traction and the effect on patient discomfort. There have been multiple studies examining the use of various distraction techniques for pain and anxiety, mainly with patients undergoing GI procedures, such as colonoscopy. The goal of our study is to investigate the use audio distraction with music from an mp3 player and headphones, and the effect on patient anxiety and pain during the placement of a skeletal traction pin. Provider-perceived patient cooperation and procedure difficulty will also be assessed.

This is a prospective randomized controlled trial at Regions Hospital in Saint Paul, MN and Jackson Memorial Hospital in Miami, Florida to compare primary outcomes of subjects between audio distraction and no audio distraction groups during traction pin placement. Recruitment of patients for inclusion in this study will be completed by the orthopedic resident placing the skeletal traction pin. Patients will be recruited for inclusion in this study after determining the medical need for placement of a skeletal traction pin. Routine care will be provided by the orthopedic resident for skeletal traction pin placement. Those included in this study and randomized into the treatment arm will be given an mp3 device and headphones to listen to a genre of music of their choosing in addition to being treated to the current routine care. Those randomized into the control arm will be treated to the current routine care without any use of music. Patients will be randomized into 2 groups; audio distraction with music versus control group with no music.

ELIGIBILITY:
Inclusion Criteria:

* Conscious, oriented, able to give informed consent
* Medical need for distal femoral or proximal tibial skeletal traction pin placement

Exclusion Criteria:

* Medical contraindication to skeletal traction
* Endotracheal intubation
* Unable to participate in verbal communication throughout the procedure and in the recovery phase
* Sensory impairment to pain
* Inability to make accurate mark on VAS 2/2 cognitive, motor or visual deficiencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Cunningham, Principal Investigator — brian.cunningham@parknicollet.com
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
In order to secure patient confidentiality and data security, all data will be de-identified. All patients will be assigned a research identification number (not their MRN) that cannot be associated with their name, birthdate, or other identifying information. Patient information will only be accessed via secure servers for Regions Hospital and on encrypted password-protected computers. If it is necessary to transmit patient data, it will be transmitted in the de-identified format, using only patient research identification numbers. At the end of the study, the electronic files will be permanently deleted and patient identifiers will be removed. All hard copies will be shredded.

REFERENCES:
- [Background] DeFroda SF, Gil JA, Born CT. Indications and anatomic landmarks for the application of lower extremity traction: a review. Eur J Trauma Emerg Surg. 2016 Dec;42(6):695-700. doi: 10.1007/s00068-016-0712-3. Epub 2016 Jul 23. PMID 27448398
- [Background] Resch S, Thorngren KG. Preoperative traction for hip fracture: a randomized comparison between skin and skeletal traction in 78 patients. Acta Orthop Scand. 1998 Jun;69(3):277-9. doi: 10.3109/17453679809000929. PMID 9703402
- [Background] Bampton P, Draper B. Effect of relaxation music on patient tolerance of gastrointestinal endoscopic procedures. J Clin Gastroenterol. 1997 Jul;25(1):343-5. doi: 10.1097/00004836-199707000-00010. PMID 9412917
- [Background] Bechtold ML, Perez RA, Puli SR, Marshall JB. Effect of music on patients undergoing outpatient colonoscopy. World J Gastroenterol. 2006 Dec 7;12(45):7309-12. doi: 10.3748/wjg.v12.i45.7309. PMID 17143946
- [Background] Palakanis KC, DeNobile JW, Sweeney WB, Blankenship CL. Effect of music therapy on state anxiety in patients undergoing flexible sigmoidoscopy. Dis Colon Rectum. 1994 May;37(5):478-81. doi: 10.1007/BF02076195. PMID 8181411
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Singer AJ, Thode HC Jr. Determination of the minimal clinically significant difference on a patient visual analog satisfaction scale. Acad Emerg Med. 1998 Oct;5(10):1007-11. doi: 10.1111/j.1553-2712.1998.tb02781.x. PMID 9862594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective randomized controlled trial was conducted to from 2018-2022 at two level-I trauma centers across North America.
Pre-assignment Details: Of the 54 enrolled participants, all 54 met inclusion criteria and were randomized into the two arms of the study.
Period: Overall Study
Arm/Group | Audio Distraction | Control
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audio Distraction | Control | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (21.8) | 52.5 (19.5) | 51.8 (20.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 14 | 17 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — kilograms per square meter (kg/m^2)
  kilograms per square meter (kg/m^2) | 27.7 (5.6) | 29.2 (11.8) | 28.5 (9.1)
Number of Participants with Substance Abuse History [Count of Participants; unit: Participants] | 7 | 4 | 11
Number of Participants with Smoking History (Yes/No) [Count of Participants; unit: Participants] | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Pain
Description: A 10-point visual analog scale for pain with 1 being the best possible outcome and 10 being the worst possible outcome. Scale is from 1-10.
Time Frame: Immediately after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Audio Distraction | Control
Number analyzed (Participants) | 28 | 26
units on a scale | 5.3 (3.2) | 6.1 (2.4)

2. Primary Outcome: Patient-reported Anxiety
Description: A 10-point visual analog scale for anxiety with 1 being the best possible outcome and 10 being the worst possible outcome. Scale is from 1-10.
Time Frame: Immediately after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Audio Distraction | Control
Number analyzed (Participants) | 28 | 26
units on a scale | 4.8 (3.3) | 7.1 (2.8)

3. Primary Outcome: Patient-reported Overall Experience
Description: A 10-point visual analog scale for patient's reported overall experience with 1 being the best possible outcome and 10 being the worst possible outcome. Scale is from 1-10.
Time Frame: Immediately after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Audio Distraction | Control
Number analyzed (Participants) | 28 | 26
units on a scale | 3.9 (2.9) | 3.5 (2.2)

4. Secondary Outcome: Procedure Time
Description: Overall time required for placement of skeletal traction pin
Time Frame: Obtained by resident from start of lidocaine injection to end of procedure (disconnecting the drill) (up to 60 minutes).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Audio Distraction | Control
Number analyzed (Participants) | 28 | 26
minutes | 16.3 (7.9) | 27.2 (17.1)

5. Secondary Outcome: Physician Reported Procedure Difficulty
Description: Resident physician will fill out survey after the procedure to evaluate the difficulty of the procedure on a 1-10 scale (1 - easy to 10- most difficult).
Time Frame: Immediately after the procedure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Audio Distraction | Control
Number analyzed (Participants) | 28 | 26
score on a scale | 2.6 (2.0) | 2.8 (1.7)

ADVERSE EVENTS:
Time Frame: Use of in-ear headphones for listening to music during the application of the traction pin which was approximately a 1-hour time frame.
Description: Only participants in the audio distraction arm who used the in-ear headphones were at risk.
Arm/Group | Audio Distraction | Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT05927480/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT05927480/ICF_001.pdf